CLINICAL TRIAL: NCT02068105
Title: A Phase 1, Randomized, Two-part Study to Evaluate the Relative Bioavailability of Two Formulations of ALKS 5461 and the Effect of Dose Titration of ALKS 5461 in Healthy Subjects
Brief Title: A Study of ALKS 5461 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-209
Record Dates: First submitted 2014-02-12; First posted 2014-02-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Pharmacokinetics
Keywords: ALKS 5461; samidorphan
MeSH Terms: interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- ALKS 5461-A (Experimental)
  Interventions: Drug: ALKS 5461
- ALKS 5461-B (Experimental)
  Interventions: Drug: ALKS 5461
- ALKS 5461 Dose 1 (Experimental)
  Interventions: Drug: ALKS 5461
- ALKS 5461 Dose 2 (Experimental)
  Interventions: Drug: ALKS 5461
- ALKS 5461 Dose 3 (Experimental)
  Interventions: Drug: ALKS 5461
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual tablet
  Arms: ALKS 5461 Dose 1; ALKS 5461 Dose 2; ALKS 5461 Dose 3; ALKS 5461-A; ALKS 5461-B
Drug: Placebo — Sublingual tablet
  Arms: Placebo

SUMMARY:
This is a study to test the safety of ALKS 5461 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Be in good physical health
* Body mass index of 18-30 kg/m2
* Agree to use an approved method of birth control for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Currently pregnant or breastfeeding
* History of or current infection with Hepatitis B Virus, Hepatitis C Virus or Human Immunodeficiency Virus (HIV)
* Current or history of any clinically significant medical or psychiatric condition
* Current abuse or dependence on alcohol or any illicit drugs
* Have used nicotine within 90 days
* Have used St. John's Wort or consumed grapefruit, grapefruit juice, or juices containing grapefruit within 30 days
* Have used any prescription or over-the-counter medication, including natural health products (with the exception of prescription birth control or hormonal replacements, acetaminophen, ibuprofen, or multivitamins) within 14 days
* Have used opioids 30 days prior to screening or have an anticipated need for opioid medication at any point during the study
* Have a history of intolerance or hypersensitivity to buprenorphine or opioid antagonists (eg, naltrexone, naloxone)
* Additional criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of ALKS 5461 treatment groups | 21 days
  The parameters for determining the bioavailability include Cmax, AUC last, and AUC(0-infinity).

SECONDARY OUTCOMES:
Safety and tolerability: Incidence of adverse events | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Randall Marshall, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Overland Park, Kansas, United States